CLINICAL TRIAL: NCT07178015
Title: Plaque-RADS Combined With Vector Flow Imaging in Assessing Carotid Atherosclerotic Risk
Brief Title: A Cohort Study on Cardiovascular and Cerebrovascular Outcomes
Status: Enrolling by invitation | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jia Liu, Clinical Professor, Sun Yat-sen University
Other Study IDs: II2025-114-02
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Atheroscleroses
MeSH Terms: conditions — Stroke; Atherosclerosis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

INTERVENTIONS:
Combination Product: ultrasound scanning — Ultrasound (US) is one of the most frequently utilized methods in carotid screening worldwide, because of its noninvasive and radiation-free nature and advantages of cost-effectiveness and convenience。

SUMMARY:
A standardized tool for grading carotid atherosclerotic plaques-dubbed Carotid Plaque-RADS (Reporting and Data System)-has recently been developed. Ultrasound (US) is one of the most frequently utilized methods in carotid screening worldwide. However, the clinical utility of US-based carotid plaque-RADS in refining stroke risk stratification beyond conventional stenosis grading has not been thoroughly validated. This study intends to conduct a bidirectional cohort study. In the retrospective part, we will collect relevant clinical data of patients and combine the Plaque-RADS scoring system to establish a risk regression prediction model for cardiovascular and cerebrovascular events in patients with carotid plaques. We will also prospectively collect a batch of patient data and incorporate ultrasound vector flow imaging and vascular hardness analysis to conduct a prospective cohort study, and further verify the accuracy and effectiveness of the model. Through this research, we aim to identify high-risk patients early, provide early intervention and treatment for high-risk individuals, and reduce the mortality and disability rates of cardiovascular and cerebrovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* patients with asymptomatic carotid plaques

Exclusion Criteria:

* suboptimal image quality or insufficiently detailed examination affecting analysis accuracy;
* recent hemorrhagic cerebral infarction, intracranial hemorrhage, or intracranial neoplasms;
* a prior history of neck radiotherapy or ipsilateral carotid artery surgical/stent procedures;
* lost to follow-up monitoring or had an estimated survival time <12 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with asymptomatic carotid plaques who underwent carotid ultrasound examinations.
Sampling Method: Non-Probability Sample
Enrollment: 855 (Estimated)
Dates: Start 2021-12-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
the occurrence of symptomatic events | 12 months after carotid ultrasound examinations

CONTACTS AND LOCATIONS:
Locations (1):
- the Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China